CLINICAL TRIAL: NCT00284388
Title: Incorporation of Muscle Qualities in Biomechanical Models of the Upper Limbs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/056
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Shoulder Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Simultaneous controlled power measurement
Procedure: Surface EMG measurement

SUMMARY:
Development of a non-invasive method for the determination of the position of optimal muscle length in the different muscles of the shoulder.

Analysis of the adaptation of the muscle to a new optimal length in patients with a shoulder prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder prosthesis

Exclusion Criteria:

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Measurement of the optimal length of the muscles of the shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be